CLINICAL TRIAL: NCT01646359
Title: Value of Pulse Pressure Variations and Corrected Flow Time in Esophageal Doppler as a Predictor of Fluid Responsiveness in Prone Position During Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-2010-0046
Record Dates: First submitted 2012-07-15; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Elective Posterior Lumbar Spinal Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- corrected flow time (Experimental)
  Interventions: Device: 1.Esophageal doppler monitor; Device: 2. philips Intelivue MP70 monitors

INTERVENTIONS:
Device: 1.Esophageal doppler monitor — 1.Esophageal doppler monitor (CARDIO Q®, DELTEX MEDICAL. Brighton, U. K.)-inserted into the esophagus and positioned approximately 35-40 cm from the teeth. The position of OED prove was confirmed by continuously measuring blood flow velocity in the descending thoracic aorta and focused to find the optimum peak velocity and waveform signal.
  Other Names: 1.CARDIO Q®, DELTEX MEDICAL. Brighton, U. K.
Device: 2. philips Intelivue MP70 monitors — 2.philips Intelivue MP70 monitors (Intellivue MP70, philips medical Systems, Suresnes, France) -a radial arterial cannula was inserted and arterial pressure waveforms were monitored through Philips Intelivue MP70 monitors. In the monitor, PPVauto was displayed in real-time. It based on automatic detection algorithms, kernel smoothing, and rank-order filters.
  Other Names: 2.intellivue MP70, philips medical Systems, Suresnes, France

SUMMARY:
In patients under mechanical ventilation, Usefulness of dynamic indices based on the heart-lung interactions for guiding volume resuscitation has been well validated. Recently, validity of pulse pressure variation (PPV) has been also reported to predict fluid responsiveness. Oesophageal Doppler (OED) allows continuous monitoring of several important hemodynamic variables. Of the OED variables, corrected flow time (FTc) has been evaluated and used as a preload index, and has been reported to predict fluid responsiveness. Prone position caused physiologic and hemodynamic changes and influenced the predictability and cut-off values of SVV and PPV for fluid responsiveness. In this prospective controlled study, the investigators evaluated the validity of PPV and FTc as predictors for fluid responsiveness in supine and prone position in patients undergoing posterior lumbar spinal fusion

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective spine surgery
* age : > 20 and < 70, 3. Patients expecting intraoperative blood loss more than 10% of estimated blood volume

Exclusion Criteria:

* arrhythmias
* BMI > 30 kg/m2
* valvular heart disease
* left ventricular ejection fraction < 50%
* history of lung disease
* pregnancy
* foreigner
* contraindications to esophageal doppler monitoring probe insertion (i.e. oesophageal stent, carcinoma of the oesophagus or pharynx, previous oesophageal surgery, oesophageal stricture, oesophageal varices, pharyngeal pouch, intra-aortic balloon pump, coarctation of the aorta, and severe coagulopathy)

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
PPV(Pulse pressure variation) | 15 minutes after induction of anaesthesia at the supine position
FTc(corrected flow time) | 15 minutes after induction of anaesthesia at the supine position

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Yang SY, Shim JK, Song Y, Seo SJ, Kwak YL. Validation of pulse pressure variation and corrected flow time as predictors of fluid responsiveness in patients in the prone position. Br J Anaesth. 2013 May;110(5):713-20. doi: 10.1093/bja/aes475. Epub 2012 Dec 28. PMID 23274783